CLINICAL TRIAL: NCT00307931
Title: Certolizumab Pegol in the Treatment of Adult Greek Patients With Moderate to Severe Crohn's Disease Who Have Been Previously Treated Successfully With Infliximab But Who Have Subsequently Lost Response or Developed Intolerance to Infliximab
Brief Title: Certolizumab Pegol for Treatment of Adult Greek Patients With Moderate to Severe Crohn's Disease Who Failed Infliximab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early because of slow recruitment
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87055; Eudract n° - 2006-002027-16
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2009-10-19 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2009-12

CONDITIONS: Crohn's Disease
Keywords: Certolizumab pegol; Cimzia; Crohn's disease; Greek patients
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab pegol (Experimental): certolizumab pegol 400 mg
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — certolizumab pegol 400 mg (lyophilized product) administered as 2 x 200 mg subcutaneous injections at Weeks 0, 2, 4, 8 and 12.
  Treatment duration: 12 weeks.
  Other Names: Cimzia

SUMMARY:
An open-label multi-center single-cohort study to assess the safety and efficacy of certolizumab pegol for the treatment of signs and symptoms of active Crohn's disease in Greek patients who have previously responded to infliximab but who no longer have a sustained response or became intolerant to infliximab

ELIGIBILITY:
Inclusion Criteria:

• Adult men and women with Crohn's disease previously responsive to infliximab who became non-responsive or intolerant

Exclusion Criteria:

* Symptomatic obstructive intestinal strictures
* Bowel resection within 4 weeks
* Current total parenteral nutrition
* Short bowel syndrome
* Concomitant disease or pathological condition that could interfere with Crohn's disease or to be harmful for the well being of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (5):
- Greece (5):
  - Heraklion, Crete
  - Athens
  - Ioannina
  - Piraeus
  - Thessaloniki

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study screened 17 subjects in 7 sites in Greece. The first subject was screened in March 2007 and the last subject was screened in February 2008. Of the 17 subjects screened, 16 were included in the Intention-to-treat population, i.e., were enrolled in the study and received at least one dose of study medication.
Groups:
- Certolizumab Pegol 400 mg: Certolizumab pegol 400 mg administered at Weeks 0, 2 ,4 ,8 and 12
Period: Overall Study
Arm/Group | Certolizumab Pegol 400 mg
Started | 16 (Number of subjects who entered the study and have been treated)
Completed | 15 (Number of subjects who completed the Week 12 visit)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 42.45 (15.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Region of Enrollment [Number; unit: participants]
  Greece | 16
Body Height [Mean (Standard Deviation); unit: cm] | 168.7 (9.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.20 (4.98)
Body Weight [Mean (Standard Deviation); unit: kg] | 64.0 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least a 100-point Decrease From Baseline in Crohn's Disease Activity Index (CDAI) Score at Week 6
Description: The CDAI score is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline, Week 6
Population: This outcome is based on the Intent-to-Treat population, defined as all subjects who were enrolled and received at least 1 dose of study medication (N=16).
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 16
participants | 7

2. Secondary Outcome: Number of Patients With at Least a 100-point Decrease From Baseline in Crohn's Disease Activity Index (CDAI) Score at Weeks 1, and 14 or Withdrawal
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, and 14 or Withdrawal
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 16
participants
  Week 1 | 6
  Week 14 or Withdrawal | 6

3. Secondary Outcome: Number of Patients With at Least a 70-point Decrease From Baseline in Crohn's Disease Activity Index (CDAI) Score at Weeks 1, 6 and 14
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, 6 and 14
Population: Due to the low number of subjects recruited only an abbreviated report was produced with limited analyses. This outcome measure was not included in the limited analyses.
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With a Crohn's Disease Activity Index (CDAI) Score ≤150 (Remission) at Weeks 1, 6 and 14 or Withdrawal
Description: as for outcome 1
Time Frame: Weeks 1, 6 and 14 or Withdrawal
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 16
participants
  Week 1 | 3
  Week 6 | 5
  Week 14 or Withdrawal | 3

5. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score at Each of Weeks 1, 2, 4, 6, 8, 12 and 14
Description: as for outcome 1
Time Frame: Weeks 1, 2, 4, 6, 8, 12 and 14
Population: as for outcome 3
Measure: Number; unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI) Score at Each of Weeks 1, 2, 4, 6, 8, 12 and 14
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, 2, 4, 6, 8, 12 and 14
Population: as for outcome 3
Measure: Number; unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: C-reactive Protein Level at Each of Weeks 1, 2, 4, 6, 8, 12 and 14
Time Frame: Weeks 1, 2, 4, 6, 8, 12 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Baseline, and Weeks 6 and 14
Description: The IBDQ Total Score is the sum of 32 responses, each ranging from 0 to 7, thus the Total Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: Baseline, and Weeks 6 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Symptoms Domain Score at Baseline, and Weeks 6 and 14
Description: The IBDQ Bowel Symptoms Domain Score is the sum of 8 responses, each ranging from 0 to 7, thus the score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: Baseline, and Weeks 6 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Symptoms Domain Score at Baseline, and Weeks 6 and 14
Description: The IBDQ Systemic Symptoms Domain Score is the sum of 8 responses, each ranging from 0 to 7, thus the score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: Baseline, and Weeks 6 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Function Domain Score at Baseline, and Weeks 6 and 14
Description: The IBDQ Emotional Function Domain Score is the sum of 8 responses, each ranging from 0 to 7, thus the score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: Baseline, and Weeks 6 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Social Function Domain Score at Baseline, and Weeks 6 and 14
Description: The IBDQ Social Function Domain Score is the sum of 8 responses, each ranging from 0 to 7, thus the score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: Baseline, and Weeks 6 and 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the treatment period and safety follow-up period, namely until 12 weeks following the last dose of study medication for each subject (which could be a time frame up to 24 weeks).
Arm/Group | Certolizumab Pegol 400 mg
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=16)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=16)
Crohn's disease (Gastrointestinal disorders) | 2 (2)
Perianal abscess (Infections and infestations) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow recruitment, namely only 17 subjects were recruited although the sample size had planned for approximately 50 subjects. As a consequence, the majority of secondary outcome measures were not summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.